CLINICAL TRIAL: NCT06012266
Title: Dose Rationale for Dapagliflozin and Empagliflozin in Paediatric Heart Failure: a Phase II.a Pharmacokinetics, Ease-of-swallow, Safety and Proof-of-concept Study Among Children 6-18 Years of Age
Brief Title: Repurposing Empagliflozin and Dapagliflozin for Paediatric Heart Failure: Translational Approach and Dose Rationale
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other); University College, London (Other)
Responsible Party: Principal Investigator, Sebastiano Lava, Principal Investigator, "Chef de clinique", Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22HL33; 2023-000441-16 (EudraCT Number)
Record Dates: First submitted 2023-08-04; First posted 2023-08-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
Keywords: child
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Intervention Model Description: Order of drug intake will be balanced and randomized, with 6 patients starting with Dapagliflozin (Visits 1-2) and subsequently switching to Empagliflozin (Visits 3-4), and 6 patients starting with Empagliflozin (Visits 1-2) and subsequently switching to Dapagliflozin (Visits 3-4).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Dapagliflozin first, Empagliflozin second (Active Comparator): Patients randomized to Group A will start with Dapagliflozin on Visit 1 and take Dapagliflozin once daily up to the day before Visit 3.
  On the day of Visit 3, they will switch to Empagliflozin once daily, to be continued up to the day preceding Visit 4.
  Interventions: Drug: Dapagliflozin tablet; Drug: Empagliflozin Tablets
- Group B: Empagliflozin first, Dapagliflozin second (Active Comparator): Patients randomized to Group B will start with Empagliflozin on Visit 1 and take Empagliflozin once daily up to the day before Visit 3.
  On the day of Visit 3, they will switch to Dapagliflozin once daily, to be continued up to the day preceding Visit 4.
  Interventions: Drug: Dapagliflozin tablet; Drug: Empagliflozin Tablets

INTERVENTIONS:
Drug: Dapagliflozin tablet — Patients randomized to Group A will start with Dapagliflozin on Visit 1 and take Dapagliflozin once daily up to the day before Visit 3.
  Patients randomized to Group B will start Dapagliflozin once daily on the day of Visit 3, to be continued up to the day preceding Visit 4.
  Dose:
  * participants ≤12 year old: 5mg once daily p.o. (commercially available tablet)
  * participants >12 year old: 10mg once daily p.o. (commercially available tablet)
Drug: Empagliflozin Tablets — Patients randomized to Group A will start with Empagliflozin on Visit 1 and take Empagliflozin once daily up to the day before Visit 3.
  Patients randomized to Group B will start Empagliflozin once daily on the day of Visit 3, to be continued up to the day preceding Visit 4.
  Dose: Empagliflozin 10mg once daily p.o. (commercially available tablet)

SUMMARY:
This study aims at exploring the use of Dapagliflozin and Empagliflozin in children and adolescents 6-18 years old with heart failure. These molecules are effective in reducing hospitalisations and mortality in adults with heart failure and are used in adolescents with type 2 diabetes mellitus, but little is known on children with heart failure. Particularly, the best dose to use in this population is currently unknown. This trial aims to:

1. define a dose rationale for this indication and age group (pharmacokinetic study),
2. assess and monitor safety,
3. assess ease-of-swallow,
4. explore middle-term (4-6 weeks) efficacy and efficacy markers.

Participants will be asked to attend 4 study visits over 4-6 weeks, and one end-study visit 2-12 weeks thereafter. Visits 1 and 3 will entail an 8h day-hospital stay, while Visits 2, 4 and the end-study visit will be outpatient clinics (approximately 2h). Participants will be asked to take the studied drug once daily during the 4-6 weeks of the study period.

All participants will take both Dapagliflozin and Empagliflozin: 6 will start with Dapagliflozin first (Visits 1-2) and then switch to Empagliflozin (Visits 3-4), while 6 will start with Empagliflozin first (Visits 1-2) and then switch to Dapagliflozin (Visits 3-4). No comparison group is foreseen for this study.

DETAILED DESCRIPTION:
Paediatric heart failure is a relevant healthcare issue, with almost 15'000 yearly hospitalizations just in the USA. Sadly, current heart failure therapy in Paediatrics is still unsatisfactory, with high in-hospital (7-26%), and 5-year mortality (30%-50%).

Among the recent improvements in adult heart failure management, impressive is the discovery that Dapagliflozin and Empagliflozin are able to reduce cardiovascular death or worsening heart failure by 25% on top of optimal medical therapy. Indeed, since 2021, they have been recommended as part of standard heart failure therapy.

In the past, paediatric heart failure trials often failed, mainly because of suboptimal dose or inappropriate formulations and endpoints.

This phase II.a, cross-over, open-label trial is designed to characterize pharmacokinetics (primary outcome), palatability, safety and explore potential efficacy markers (secondary outcomes) of Dapagliflozin and Empagliflozin in 12 heart failure children, so to inform the design and performance of subsequent, state-of-the-art, high-quality efficacy trials.

Participants will first receive Drug A (either Dapagliflozin, n=6, or Empagliflozin, n=6) during 3-5 weeks, followed by the other molecule (Drug B) for 2 weeks. They will have 4 visits, one end-study visit and 11-15 pharmacokinetic samples (depending on their weight). The timing of these samples will be optimized exploiting contemporary modeling and simulation techniques.

Safety evaluation will occur throughout the study, while palatability will be evaluated at Visits 1 (Drug A) and 3 (Dug B), and efficacy markers at Visits 1, 3 and 4.

Pharmacokinetic modeling will characterize primary and secondary pharmacokinetic parameters and allow to define the optimal paediatric dose, informing both current compassionate-care use and the design of future efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 18 years of age, followed either as in- or outpatients at the Heart failure unit, Great Ormond Street Hospital NHS Foundation Trust, London or at the Paediatric Cardiology Unit, Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne University Hospital, Lausanne, Switzerland will be eligible for inclusion.
* Currently on heart failure medication (any drug or any combination).
* Patients should potentially benefit from adding a SGLT2i (as judged by the treating physician and the local PI or Co-PI).
* Patients need to be on stable medical treatment, defined as no new heart failure drug started over the preceding 2 weeks and no major drug dose modification (apart minor adaptations, like weight adaptations, rounding or formulation changes) during the 2 weeks prior to enrolment.
* Adolescents, respectively parents or caregivers of children, capable of giving informed consent.

Exclusion Criteria:

* Inability to understand and go through the informed consent procedure.
* Inability to receive medications per os or through a nasogastric tube.
* Patients on either Insulin or Metformin will be excluded from participation. This implies the exclusion of patients with Diabetes mellitus (either type 1 or type 2 or other rare forms) necessitating either insulin or metformin.
* Type 1 Diabetes mellitus or any underlying metabolic disease associated with hypoglycaemias.
* Body weight <13kg.
* Current smokers (defined as >1 cigarette/week).
* Use of any other nicotine-delivering product (e.g. nicotine patches).
* Any known illicit drug abuse.
* Active chronic HBV, HCV or HIV.
* Any major surgery within 4 weeks of first dose administration.
* Blood transfusion recipient within 4 weeks of dose administration.
* eGFR =<45mL/min/1.73m2 (simplified Schwartz formula).
* K+ >6.5mmol/L.
* Blood glucose <4mmol/L.
* There are no blood pressure exclusion criteria foreseen, but participants need to be haemodynamically stable, as assessed by the local investigator (board-certified paediatric cardiologist).
* Sustained or symptomatic arrhythmia insufficiently controlled with drug and/or device therapy.
* Cardio-surgical procedure within the 2 months prior to Visit 1, or interventional cardiac catheterization within 2 weeks prior to Visit 1, or the patient is planned to undergo cardiac surgery or an interventional cardiac catheterization during the study period (i.e. in the 6 weeks following Visit 1).
* Post-menarchal female patients of childbearing potential cannot be included.
* Known lactose intolerance, galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
* Known allergies to excipients of either Dapagliflozin or Empagliflozin.
* Significant medical history of active severe medical disease.
* Significant liver disease, Child Pugh Class C, or significant laboratory abnormalities at enrolment.
* Significant gastroenterological or hepatic disease that could significantly impair absorption or metabolism of orally administered drugs.
* Any medical co-morbidity, which is deemed incompatible (or only with relevant risk) with study participation by the treating clinician and/or the study investigator.
* Active urinary tract infection (being treated with antibiotics at the moment of Visit 1) or other relevant bacterial infection, as judged by the treating clinician and/or the study investigator.
* The patient is currently participating in another interventional clinical trial or has participated in such a trial during the <14 days before Visit 1 (or if enrolment in this study is incompatible with the protocol of that preceding trial).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics 1: Dapagliflozin, respectively Empagliflozin half-life | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  This will be derived by pharmacokinetic analysis and modeling, basing on Dapagliflozin, respectively Empagliflozin, concentrations at the different time-points (5-6 samples [according to weight] at Visit 1, 1 opportunistic sample at Visits 2 and 3 for Drug A; 5-6 samples [according to weight] at Visit 3 and 1 opportunistic sample at Visit 4 for Drug B; the timing of the samples will be optimized with modeling & simulation techniques).
Pharmacokinetics 2: Dapagliflozin, respectively Empagliflozin Volume of distribution | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  This will be derived by pharmacokinetic analysis and modeling, basing on Dapagliflozin, respectively Empagliflozin, concentrations at the different time-points (5-6 samples [according to weight] at Visit 1, 1 opportunistic sample at Visits 2 and 3 for Drug A; 5-6 samples [according to weight] at Visit 3 and 1 opportunistic sample at Visit 4 for Drug B; the timing of the samples will be optimized with modeling & simulation techniques).
Pharmacokinetics 3: Dapagliflozin, respectively Empagliflozin AUC | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  This will be derived by pharmacokinetic analysis and modeling, basing on Dapagliflozin, respectively Empagliflozin, concentrations at the different time-points (5-6 samples [according to weight] at Visit 1, 1 opportunistic sample at Visits 2 and 3 for Drug A; 5-6 samples [according to weight] at Visit 3 and 1 opportunistic sample at Visit 4 for Drug B; the timing of the samples will be optimized with modeling & simulation techniques).

SECONDARY OUTCOMES:
Safety 1 - eGFR | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  Creatinine (respectively Cystatin C in DMD participants) will be collected in order to calculate eGFR (bedside Schwartz formula, respectively Filler equation).
Safety 2 - Occurrence of hypoglycemia | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  Blood glucose will be checked three times at Visit 1 and Visit 3 (baseline, at the time of 2nd PK sampling, which will be individualized but will be at approximately 2-3h post-intake, and before discharge at 8h post-intake), as well as once at Visits 2 and 4 (together with PK sampling). Outcome measure: number of patients experiencing hypoglycemia.
Safety 3 - Occurrence of ketoacidosis | Visits 1-4 (Visit 1 = day 1, Visit 2 = week 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  The outcome is presence (or absence) of ketoacidosis. This will be assessed at Visits 1, 2, 3, and 4. Outcome measure: number of patients experiencing ketoacidosis.
Ease-of-swallow | Visit 1, Visit 3 (Visit 1 = day 1, Visit 3 = week 3 to 5 after study start)
  Ease of swallow will be assessed by means of facial hedonic scales, according to our standard procedure, at Visit 1 (Drug A), and Visit 3 (Drug B). (Scale 1 to 4, 1 being the worse and 4 the best score: very difficult - difficult - possible - easy to swallow.)
Efficacy and efficacy markers (exploratory) 1 - Heart failure severity class | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  Symptoms, clinical signs, NYHA (if >8 years of age) / Ross (if <8 years of age) class assignment. NYHA and Ross heart failure classes share the same scale of I (no limitation of physical activity) to IV (symptoms at rest). Analysis will be performed at Visit 1, Visit 3 and Visit 4. Outcome: change between Visit 1 and Visit 4.
Efficacy and efficacy markers (exploratory) 2 - NT-proBNP level | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  Analysis will be performed at Visits 1, 3 and 4. Outcome: change between Visit 1 and Visit 4.
Efficacy and efficacy markers (exploratory) 3 - Echocardiography 1: Left-ventricular end-diastolic diameter (LVEDd) | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  LVEDd (mm) will be measured at Visits 1, 3 and 4. Outcome: change between Visit 1 and Visit 4.
Efficacy and efficacy markers (exploratory) 4 - Echocardiography 2: Left-ventricular end-systolic diameter (LVESd) | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  LVESd (mm) will be measured at Visits 1, 3 and 4. Outcome: change between Visit 1 and Visit 4.
Efficacy and efficacy markers (exploratory) 5 - Echocardiography 3: Fractional shortening (FS) | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  FS (%) will be measured at Visits 1, 3 and 4. Outcome: change between Visit 1 and Visit 4.
Efficacy and efficacy markers (exploratory) 6 - Echocardiography 4: Left ventricular ejection fraction (LV-EF) | Visits 1, 3 and 4 (Visit 1 = day 1, Visit 3 = week 3 to 5, Visit 4 = week 4 to 6 after study start)
  LV-EF (%) will be measured at Visits 1, 3 and 4. Outcome: change between Visit 1 and Visit 4.

OTHER OUTCOMES:
Efficacy markers (exploratory), Mechanistic insights - 1: body weight (kg) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on fluid status, body weight will be assessed (outcome: change between Visit 1 and Visit 4).
Efficacy markers (exploratory), Mechanistic insights - 2: heart rate (bpm) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on sympathetic activation, heart rate (in bpm) will be assessed (outcome: change between Visit 1 and Visit 4).
Efficacy markers (exploratory), Mechanistic insights - 3: blood pressure (SBP/DBP, mmHg) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on sympathetic activation, blood pressure (SBP and DBP, in mmHg) will be assessed (outcome: change between Visit 1 and Visit 4).
Efficacy markers (exploratory), Mechanistic insights - 4: b-hydroxybutyrate (mmol/L) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on metabolism shift, b-hydroxybutyrate will be assessed (outcome: change between Visit 1 and Visit 4).
Efficacy markers (exploratory), Mechanistic insights - 5: haemoglobin (g/L) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on haemoglobin, haemoglobin will be assessed (outcome: change between Visit 1 and Visit 4).
Efficacy markers (exploratory), Mechanistic insights - 6: uric acid (mmol/L) | Visit 1, Visit 4 (Visit 1 = day 1, Visit 4 = week 4 to 6 after study start)
  To explore the effect of SGLT2 inhibitors on uric acid homeostasis, uric acid will be assessed (outcome: change between Visit 1 and Visit 4).

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano A.G. Lava, MD MSc, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
Locations (3):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland
- United Kingdom (2):
  - University College London, London, Greater London
  - Great Ormond Street Hospital NHS Foundation Trust, London, Greater London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Das BB. Current State of Pediatric Heart Failure. Children (Basel). 2018 Jun 28;5(7):88. doi: 10.3390/children5070088. PMID 29958420
- [Background] Rossano JW, Kim JJ, Decker JA, Price JF, Zafar F, Graves DE, Morales DL, Heinle JS, Bozkurt B, Towbin JA, Denfield SW, Dreyer WJ, Jefferies JL. Prevalence, morbidity, and mortality of heart failure-related hospitalizations in children in the United States: a population-based study. J Card Fail. 2012 Jun;18(6):459-70. doi: 10.1016/j.cardfail.2012.03.001. Epub 2012 Apr 10. PMID 22633303
- [Background] Ahmed H, VanderPluym C. Medical management of pediatric heart failure. Cardiovasc Diagn Ther. 2021 Feb;11(1):323-335. doi: 10.21037/cdt-20-358. PMID 33708503
- [Background] Andrews RE, Fenton MJ, Dominguez T, Burch M; British Congenital Cardiac Association. Heart failure from heart muscle disease in childhood: a 5-10 year follow-up study in the UK and Ireland. ESC Heart Fail. 2016 Jun;3(2):107-114. doi: 10.1002/ehf2.12082. Epub 2016 Jan 24. PMID 27812385
- [Background] Newland DM, Law YM, Albers EL, Friedland-Little JM, Ahmed H, Kemna MS, Hong BJ. Early Clinical Experience with Dapagliflozin in Children with Heart Failure. Pediatr Cardiol. 2023 Jan;44(1):146-152. doi: 10.1007/s00246-022-02983-0. Epub 2022 Aug 10. PMID 35948644
- [Background] Towbin JA, Lowe AM, Colan SD, Sleeper LA, Orav EJ, Clunie S, Messere J, Cox GF, Lurie PR, Hsu D, Canter C, Wilkinson JD, Lipshultz SE. Incidence, causes, and outcomes of dilated cardiomyopathy in children. JAMA. 2006 Oct 18;296(15):1867-76. doi: 10.1001/jama.296.15.1867. PMID 17047217
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Cella M, Knibbe C, Danhof M, Della Pasqua O. What is the right dose for children? Br J Clin Pharmacol. 2010 Oct;70(4):597-603. doi: 10.1111/j.1365-2125.2009.03591.x. No abstract available. PMID 21087295
- [Background] Benjamin DK Jr, Smith PB, Jadhav P, Gobburu JV, Murphy MD, Hasselblad V, Baker-Smith C, Califf RM, Li JS. Pediatric antihypertensive trial failures: analysis of end points and dose range. Hypertension. 2008 Apr;51(4):834-40. doi: 10.1161/HYPERTENSIONAHA.107.108886. Epub 2008 Mar 10. PMID 18332283
- [Background] European Union. Ethical considerations for clinical trials on medicinal products conducted with the paediatric population. Eur J Health Law. 2008 Jul;15(2):223-50. doi: 10.1163/157180908x333228. PMID 18988606
- [Background] Bellanti F, Della Pasqua O. Modelling and simulation as research tools in paediatric drug development. Eur J Clin Pharmacol. 2011 May;67 Suppl 1(Suppl 1):75-86. doi: 10.1007/s00228-010-0974-3. Epub 2011 Jan 19. PMID 21246352
- [Background] Bellanti F, Di Iorio VL, Danhof M, Della Pasqua O. Sampling Optimization in Pharmacokinetic Bridging Studies: Example of the Use of Deferiprone in Children With beta-Thalassemia. J Clin Pharmacol. 2016 Sep;56(9):1094-103. doi: 10.1002/jcph.708. Epub 2016 Apr 1. PMID 26785826
- [Background] Lava SA, Simonetti GD, Bianchetti AA, Ferrarini A, Bianchetti MG. Prevention of vitamin D insufficiency in Switzerland: a never-ending story. Int J Pharm. 2013 Nov 30;457(1):353-6. doi: 10.1016/j.ijpharm.2013.08.068. No abstract available. PMID 24216246
- [Background] Braunwald E. Gliflozins in the Management of Cardiovascular Disease. N Engl J Med. 2022 May 26;386(21):2024-2034. doi: 10.1056/NEJMra2115011. No abstract available. PMID 35613023
- [Background] Zelniker TA, Braunwald E. Mechanisms of Cardiorenal Effects of Sodium-Glucose Cotransporter 2 Inhibitors: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Feb 4;75(4):422-434. doi: 10.1016/j.jacc.2019.11.031. PMID 32000955
- [Background] Joshi SS, Singh T, Newby DE, Singh J. Sodium-glucose co-transporter 2 inhibitor therapy: mechanisms of action in heart failure. Heart. 2021 Jun 11;107(13):1032-1038. doi: 10.1136/heartjnl-2020-318060. PMID 33637556